CLINICAL TRIAL: NCT00281476
Title: The Effect of High Dose Simvastatine on Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vejle Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-004933-16
Record Dates: First submitted 2006-01-23; First posted 2006-01-24 (Estimated); Last update posted 2011-11-01 (Estimated); Status verified 2011-10

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; statins; bone
MeSH Terms: conditions — Multiple Myeloma | interventions — Simvastatin

INTERVENTIONS:
Drug: Simvastatine

SUMMARY:
The purpose of the study is to evaluate the effect of high doses of Simvastatine on bone metabolisme and biochemical markers of disease in Multiple Myeloma

ELIGIBILITY:
Inclusion Criteria:

* multiple myeloma-patients in need of treatment
* stable og progressive disease
* age = or > 18 years
* performance status < 3
* life expectancy > 3 months

Exclusion Criteria:

* pregnancy
* patients incapable of giving personally concent
* renal insufficiens with creatinine clearance below 25 ml/min
* alanin aminotransferasis > 2,5 x upper reference limit
* thyroxine below lower reference limit
* known familiar muscle-disease ar previous myopati
* creatinine kinase > 10 x upper reference limit
* medication with drugs with known interactions wiht simvastatine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2006-02; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Response estimated by internationally approved criteria after 8 weeks of intermittend treatment with simvastatine | 8 weeks after treatment start

SECONDARY OUTCOMES:
Changes in markers of bone metabolisme after 8 weeks of intermittend treatment with simvastatine | 8 weeks after start of treatment
Toxicity according to CTC after 8 weeks of intermittend treatment with simvastatine | 8 weeks after start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Torben Plesner, DMSc., Principal Investigator